CLINICAL TRIAL: NCT06668324
Title: Multiple Sclerosis Patient Experience on Kesimpta and Ocrevus Subcutaneous Formulation (MS-PEKOS)
Brief Title: Multiple Sclerosis Patient Experience on Kesimpta and Ocrevus Subcutaneous Formulation
Acronym: MS-PEKOS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157AUS25
Record Dates: First submitted 2024-10-22; First posted 2024-10-31 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ofatumumab
- ocrelizumab SC formulation

SUMMARY:
The study aims to compare the experiences, including injection-related reactions (IRRs) of patients newly receiving ofatumumab to those starting to receive ocrelizumab SC formulation

ELIGIBILITY:
Inclusion Criteria:

1. Ability to use a mobile device or computer with broadband internet access (or data streaming available)
2. Ability to read, understand, and respond in English
3. Adult aged 18 years of age or over at the time of the survey
4. Self-confirmed diagnosis of MS
5. Prescribed either OMB or OCR SC and will receive their first injection (Day 0) followed by completing the study survey between Day 1 and Day 7

Exclusion Criteria:

1. Participated in an OMB or OCR randomized clinical trial
2. Previously treated with OMB or OCR SC
3. Cognitive impairment that impacts the patient's ability to participate in a survey study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MS who are prescribed and initiating OMB or OCR SC and who are living in the US at the time of the survey will be invited to participate following a referral from their healthcare providers
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reported local injection-related reaction post first injection | Day 1- 7 post first injection, at the time of survey completion
  Proportion of patients reported local injection-related reactions (including pain, erythema, induration, and pruritus) by using modified Defense and Veterans Pain Rating Scale (DVPRS)

SECONDARY OUTCOMES:
Proportion of patients in a 5-Likert scale for satisfaction on injection-related experience (post first injection) | Day 1 - 7 post first injection, at the time of survey completion
  Proportion of patients in a 5-Likert scale (extremely dissatisfied, dissatisfied, neutral, satisfied, and extremely satisfied) for satisfaction on injection-related experience
Proportion of patients reported local injection-related reaction post second injection | Day 1- 7 post second injection, at the time of survey completion
  Proportion of patients reported local injection-related reactions (including pain, erythema, induration, and pruritus) by using modified Defense and Veterans Pain Rating Scale (DVPRS)
Proportion of patients in a 5-Likert scale for satisfaction on injection-related experience (post second injection) | Day 1- 7 post second injection, at the time of survey completion
  Proportion of patients in a 5-Likert scale (extremely dissatisfied, dissatisfied, neutral, satisfied, and extremely satisfied) for satisfaction on injection-related experience

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No